CLINICAL TRIAL: NCT00201084
Title: Physician Uncertainty Reduction for Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); The University of Texas Health Science Center, Houston (Other); Kelsey Research Foundation (Other)
Responsible Party: Principal Investigator, David Hyman, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276; R01HL078589 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Uncertainty reduction tools, at physician discretion, 24 hour ambulatory BP monitoring and/or electronic bottle cap monitoring and/or lifestyle counseling
  Interventions: Behavioral: Uncertainty reduction
- 2 (No Intervention): Usual primary care

INTERVENTIONS:
Behavioral: Uncertainty reduction — At physician discretion, 24 hour ambulatory BP monitoring and/or electronic bottle cap monitoring and/or lifestyle counseling
  Arms: 1

SUMMARY:
The purpose of this study is to test the theory that a major factor in poor blood pressure (BP) control is that physicians fail to intensify antihypertensive therapy for their patients.

DETAILED DESCRIPTION:
BACKGROUND:

A large amount of literature suggests that the majority of "uncontrolled" hypertensives are under medical care, and that lack of control is largely explained by physicians not intensifying treatment to achieve the BP targets recommended in the national guidelines. Traditional physician education, feedback, and reminders have a limited effect in promoting a rapid rate of guideline implementation. The theoretical framework of diffusion of innovations suggests that providing physicians with tools to reduce uncertainty about the attributes of a guideline may accelerate the adoption process. The presumed barriers to treatment intensification for uncontrolled hypertension are: 1) uncertainty over the patient's "true" BP; 2) uncertainty over whether the patient is adherent to medications already prescribed; and 3) uncertainty over the benefits of adding medications when patients express preference for lifestyle modification.

DESIGN NARRATIVE:

This cluster randomized trial in 10 primary care clinics (5 intervention and 5 control) will test the hypothesis that an intervention based on diffusion of innovations theory, and targeting provider treatment actions, will increase the prevalence of BP control to Joint National Committee-7(JNC-7) recommended levels in African American patients (greater than 140/90 mm Hg or greater 130/80 mm Hg if the patient has diabetes). The uncertainty reduction tools in the "Uncertainty Reduction to Accelerate Diffusion (URAD)" practices will include: 24-hour ambulatory BP monitoring, electronic bottle-cap monitoring of medication adherence, and medication and lifestyle counseling. The "Usual Practice (UP)" physicians will receive education about the guidelines and a "placebo" chart form indicating the patient is being followed in a BP control study. The 10 participating clinics represent a large, multi-site private group practice and a public health care system. Sixty-seven patients per clinic (670 total) will be enrolled when the intervention is initiated, and their BP and self-reported medication and lifestyle adherence will be monitored for two years. Sixty percent of the sample will be African American, and the study will have 90% power to detect a difference of 20% in the prevalence of hypertension control in the African Americans as a result of the intervention (50% control in URAD clinics vs. 30% control UP clinics). Secondary endpoints will include BP measurements by study staff under standardized conditions, physician treatment intensification actions, patient adherence, characteristics of doctor-patient communication associated with treatment action, use of the URAD components, and physician knowledge and beliefs about the JNC 7 guidelines and their relationship to BP control. Analysis of secondary endpoints will include race. The research team has collaborated with both health systems in previous studies, and is experienced in conducting hypertension control and behavioral intervention studies in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Kept appointment on index visit day (see patient sampling and recruitment methods below)
* Had one previous visit to the setting within the past year and identified the setting as his/her usual source of care
* Average clinic BP on index visit and one most recent previous visit was equal to or greater than 140 mm Hg systolic or 90 mm Hg diastolic (130/80 mm Hg if diabetic)
* Acknowledges understanding of the study goals and methods and gives informed consent to participate in study measurements and other procedures

Exclusion Criteria:

* Cognitive or other functional impairment sufficient to limit patient's ability to give informed consent, keep follow-up appointments, and participate actively in adherence to his or her treatment regimen
* Renal insufficiencies or renal failure based on a recent serum creatinine greater than 2.0 or chart diagnosis
* Planning to leave the Houston area within the next two years
* Severe, life-threatening illness that makes hypertension treatment a secondary priority

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Expressed as the proportion of patients with average clinic BP less than 140/90 mm Hg in the previous two visits (130/80 mm Hg if the patient also has diabetes) | 24 months

SECONDARY OUTCOMES:
Actual measure clinic systolic and diastolic BP, patient physician communication patterns | 24 months
Patient adherence to medication and healthy lifestyle | 24 months
Physician knowledge, attitude, and beliefs about JNC-7 goals and barriers to achievement of the treatment goals and cost | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David J. Hyman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Pavlik VN, Greisinger AJ, Pool J, Haidet P, Hyman DJ. Does reducing physician uncertainty improve hypertension control?: rationale and methods. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):257-63. doi: 10.1161/CIRCOUTCOMES.109.849984. PMID 20031846
- [Result] Grigoryan L, Pavlik VN, Hyman DJ. Characteristics, drug combinations and dosages of primary care patients with uncontrolled ambulatory blood pressure and high medication adherence. J Am Soc Hypertens. 2013 Nov-Dec;7(6):471-6. doi: 10.1016/j.jash.2013.06.004. Epub 2013 Jul 23. PMID 23890931
- [Result] Grigoryan L, Pavlik VN, Hyman DJ. Predictors of antihypertensive medication adherence in two urban health-care systems. Am J Hypertens. 2012 Jul;25(7):735-8. doi: 10.1038/ajh.2012.30. Epub 2012 Mar 22. PMID 22441507
- [Result] Hyman DJ, Pavlik VN, Greisinger AJ, Chan W, Bayona J, Mansyur C, Simms V, Pool J. Effect of a physician uncertainty reduction intervention on blood pressure in uncontrolled hypertensives--a cluster randomized trial. J Gen Intern Med. 2012 Apr;27(4):413-9. doi: 10.1007/s11606-011-1888-1. Epub 2011 Oct 27. PMID 22033742